CLINICAL TRIAL: NCT06363175
Title: Patient-Reported Experience Measures in Vascular Surgery Enhancement Study
Brief Title: PREMs In Vascular SurgERy Enhancement Study
Acronym: PREMIERE
Status: Not yet recruiting | Type: Observational
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: Welsh Value in Health Centre (WViHC) (Unknown); Centre for Healthcare Evaluation, Device Assessment, and Research (CEDAR) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 8737; 343073 (Other: Integrated Research Application system (IRAS))
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Vascular Diseases; Patient Empowerment; Patient Satisfaction; Patient Engagement; Surgery
Keywords: Patient Reported Experience Measure; PREM; Vascular surgery; Patient centred care
MeSH Terms: conditions — Vascular Diseases; Patient Participation; Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
THE PROBLEM:

Patient Reported Experience Measures (PREMs) ask patients about their healthcare service experience. It gives them a voice to share their views. PREMs allow healthcare providers (HCPs) to see where care is good, and where they could improve. Vascular surgery is a surgical speciality looking after people's blood vessels (arteries and veins).

There is no PREM available for vascular patients. The research team want to create a PREM for this patient group.

WHY IT IS IMPORTANT:

A PREM allows HCPs to record and understand patients' experiences of their treatment. It gives patients a way to provide feedback on their healthcare experience. PREMs can help HCPs make changes to patients' care, identifying areas of good practice and areas for improvement. The Welsh Government is keen to support the use of PREMs.

AIMS:

To develop a PREM specific to vascular surgery patients.

RESEARCH PLAN:

The research team will summarise the literature about PREMs in surgery. The research team will then run focus groups and interviews with patients and staff to create a 'draft' PREM for vascular patients in Wales. The 'draft' PREM will be translated into Welsh.

In the second phase, a larger number of vascular patients (100-300 depending on how long the 'draft' PREM is) from hospitals across Wales will complete the questionnaire. Statistical tests will look at the results to see if the questionnaire works well to capture patients' experiences. Based on these results, small changes will be made to make the 'draft' PREM better. This will make sure the 'final PREM' is ready for widespread use in Wales and beyond.

PATIENT AND PUBLIC INVOLVEMENT:

The patients' experience team at CAVUHB has reviewed our patients' materials. Our research team includes PPI co-applicants (DC and AH). DC a double amputee who has had many vascular operations. DC has experience raising awareness about vascular disease through public forums like the Limbless Association Charity and BBC Radio Wales. AH has issues with her leg due to smoking and had a keyhole operation to help with that. She had some problems after the procedure This is her first time as a PPI representative. DC and AH supported our research design and will be steering group members. Also, our research focuses on giving patients a voice and will include patients across Wales. A diverse group of patients will be involved across all stages of the PREM development.

DETAILED DESCRIPTION:
Background: PREMs have emerged as instruments designed to capture patients' experiences of their healthcare journey. No PREMs have been developed or validated to be used among vascular surgery patients specifically.

Objectives: To develop and validate a PREM specific to vascular surgery, assessing the patient's experience and satisfaction with their care and treatment.

Study design and methods: Patient Reported Experience Measures In Vascular Surgery Enhancement Study (PREMIERE) is a multi-site sequential mixed-methods cohort design, incorporating qualitative and quantitative approaches in two phases. The first phase will focus on developing a draft PREM for vascular surgery patients, while the second phase will aim to validate the draft PREM to create a 'final PREM'. Patient inclusion criteria are: (i) age ≥18 ; (ii) have undergone a vascular procedure (iii) experienced an inpatient vascular care within the previous 3 months; (iv) not cognitively impaired; (v) willing and able to provide written consent for participation; (vi) able to communicate in English or Welsh.

Statistical analysis: For the qualitative phase, inductive thematic analysis will be carried out using the non-numerical data analysis for Windows software NVivo . For quantitative data, psychometric tests such as item analysis, internal consistency, construct validity, and principal component analysis with varimax rotation will be used to extract factors. Quantitative data will be analysed using IBM SPSS Statistics (Version 27) software.

Anticipated impact: PREMIERE will contribute to the development of a robust and context-specific PREM for vascular patients. This PREM will provide a valuable tool for assessing and improving the in-patient vascular surgery pathway, including pre-operative, peri-operative, and post-operative phases. Also, the utilization of a robust vascular PREM presents a transformative opportunity to benchmark and enhance the performance of vascular units.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have recently (within the last three months) undergone a vascular procedure or intervention under the care of a vascular surgery team in the inpatient setting.
* Adults aged 18 years or older
* Not cognitively impaired (as determined by medical reports and/or self-reporting).
* Willing and able to provide written consent for participation.
* Able to speak, read and write English or Welsh

Exclusion Criteria:

* Patients who lack capacity or suffer from cognitive impairment.
* Patients who are unable to speak, read and write English or Welsh.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing in-patient vascular care, which involves specialized vascular surgery for hospital-admitted individuals, including those recently discharged with conditions like peripheral artery disease. Recruitment will engage patients preoperatively and post-service (within 1-3 months) to minimize bias. The study will target UK's central vascular units for diverse patient demographics. Consistent eligibility criteria will apply to both study phases (development and validation).
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Degree of Validity of the PREM | Day 0, Day 30
  Validity: The extent to which a measure assesses what it intends to measure.
Degree of Reliability of the PREM | Day 0, Day 30
  Reliability: The consistency and stability of a measure over time and across different conditions.
Degree of Responsiveness of the PREM | Day 0, Day 30
  Responsiveness: The ability of a measure to detect change over time in the concept being measured.
Degree of Feasibility of implementing the PREM in clinical practice | Day 0, Day 30
  Feasibility: The practicality and suitability of implementing a measure in a specific setting or context.

CONTACTS AND LOCATIONS:
Overall Officials: David C Bosanquet, FRCS, Principal Investigator — CARDIFF & VALE UNIVERSITY LHB
Locations (1):
- Southeast Wales Vascular Network-Cardiff and Vale University Health Board, Cardiff, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The full dataset is not expected to be made available for secondary research. In accordance with standard measures to prevent statistical disclosure, quantitative data relating to five or fewer individuals will be aggregated or redacted prior to publication. Similarly, full focus group transcripts will not be made available to external individuals or organisations due to the possibility of statistical disclosure from these qualitative data.

REFERENCES:
- [Derived] Darwish M, Palmer R, Coulson J, Bosanquet DC, Withers K. Patient-Reported Experience Measures in Vascular Surgery Enhancement (PREMIERE) study: protocol for a mixed-methods study to develop and validate a vascular surgery-specific patient-reported experience measure. BMJ Open. 2025 Jul 5;15(7):e089240. doi: 10.1136/bmjopen-2024-089240. PMID 40617619